CLINICAL TRIAL: NCT02256982
Title: A Pilot Study of Neoadjuvant Therapy With Gemcitabine and Cisplatin in Patients With Resectable or Unresectable Intrahepatic Cholangiocarcinoma
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow accrual.
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Theodore Sunki Hong, Principal Investigator, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-275
Record Dates: First submitted 2014-09-25; First posted 2014-10-06 (Estimated); Results first posted 2016-04-13 (Estimated); Last update posted 2016-04-13 (Estimated); Status verified 2016-04

CONDITIONS: Unresectable Intrahepatic Cholangiocarcinoma; Resectable Intrahepatic Cholangiocarcinoma
Keywords: unresectable intrahepatic cholangiocarcinoma; resectable intrahepatic cholangiocarcinoma
MeSH Terms: interventions — Gemcitabine; Cisplatin; Surgical Procedures, Operative; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Resectable Disease (Experimental): * Consent and Registration
  * 3 cycles of gemcitabine + cisplatin
  * Evaluate for surgery* (weeks 10-15)
    -- Patients who are eligible for surgery at restaging will receive surgery; patients not eligible for surgery at restaging will receive radiation therapy.
  * Proceed to surgery
  * Additional care as recommended; may include additional cycles of GEM + CDDP on a 21 day cycle and/or post-op radiation as recommended by treating medical oncologist and radiation oncologist
  Interventions: Drug: Gemcitabine; Drug: Cisplatin; Procedure: Surgery
- Unresectable Disease (Experimental): * Consent and Registration
  * 3 cycles of gemcitabine + cisplatin
  * Evaluate for surgery* (weeks 10-15)
  * Patients who are eligible for surgery at restaging will receive surgery; patients not eligible for surgery at restaging will receive radiation therapy.
  * Proceed to radiation therapy with protons or photons, determined by available resources
  * Additional cycles of GEM + CDDP on a 21 day cycle as recommended by treating medical oncologist
  Interventions: Drug: Gemcitabine; Drug: Cisplatin; Radiation: Radiation

INTERVENTIONS:
Drug: Gemcitabine
  Other Names: Gemzar
Drug: Cisplatin
  Other Names: Platinol®; Platinol-AQ®; cis-DDP; cis-Platinum II; cis-Diamminedichloroplatinum; DDP
Procedure: Surgery — Surgical Resection and Lymphadenectomy
  Arms: Resectable Disease
Radiation: Radiation — Radiation Therapy
  Arms: Unresectable Disease

SUMMARY:
This research study is evaluating the use of radiation therapy in combination with chemotherapy as a possible treatment for intrahepatic cholangiocarcinoma, a rare form of gastrointestinal cancer.

DETAILED DESCRIPTION:
This study is to assess the possibility of using radiation therapy to treat intrahepatic cholangiocarcinoma. Radiation therapy is used for many other types of malignancies, but its use for the treatment of this form of gastrointestinal cancer has been limited. This treatment is still being studied as research doctors are trying to find out more about its use in the treatment of your form of gastrointestinal cancer. Short course photon radiation and short course proton beam radiation therapies are FDA (U.S. Food and Drug Administration) approved radiation delivery systems. This study will also test the safety of neoadjuvant chemotherapy versus adjuvant chemotherapy. Neoadjuvant therapy is treatment given as a first step to shrink a tumor before the main treatment, which is usually surgery, is given. Adjuvant therapy is additional cancer treatment given after the primary treatment to lower the risk that the cancer will come back.

The current standard of care for patients with intrahepatic cholangiocarcinoma is to offer surgical resection to all patients who have resectable disease and are able to tolerate a major surgical intervention.

The study interventions involved this trial may include one or more of the following:

* Chemotherapy (Gemcitabine and Cisplatin)
* Surgical Resection and Lymphadenectomy
* Radiation Therapy

ELIGIBILITY:
Inclusion Criteria:

* Participants must meet the following criteria on screening examination to be eligible to participate in the study:
* Participants must have histologically confirmed Intrahepatic Cholangiocarcinoma (IHC) without evidence of extrahepatic metastasis.
* Participants must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥ 20 mm with conventional techniques or as ≥10 mm with spiral CT scan.
* Participants with resectable disease must have a single tumor (with no satellite lesions) with a total diameter or longest dimension of ≤ 20cm. Patients with unresectable disease must have a total tumor diameter of <20cm and ≤ 3 lesions. Satellite lesions defined as lesions ≤ 2cm from the dominant lesion are permitted for participants with unresectable disease
* Patients are not allowed to receive prior surgery or chemotherapy for the IHC.
* Patients with age ≥18 will be included in the study.
* Expected survival must be three months or greater.
* ECOG performance status ≤ 2 (Karnofsky ≥ 70%, see Appendix A).
* Participants must have normal organ and marrow function as defined below:

  * Absolute neutrophil count ≥ 1,500/mcL
  * Platelets ≥ 100,000/mcL
  * Total bilirubin ≤ 2.5 mg/dl
  * AST (SGOT)/ALT (SGPT) ≤ 5.0 X institutional upper limit of normal
  * Creatinine within normal institutional limits or creatinine clearance ≥ 60 mL/min/1.73 m2 for subjects with creatinine levels above institutional normal .
* No other known active secondary primary malignancy.
* If patient has underlying cirrhosis, only Child-Pugh classification Group A patients may be included in the resectable cohort of this study. For patients with unresectable disease, Child-Pugh classification Groups A and B are allowed. Clinical assessment of ascites and encephalopathy is required. Child-Pugh classification must be determined for all study participants at the time of eligibility analysis. Note albumin and PT/INR are required for Child-Pugh classification; these labs should be drawn with the other labs required for eligibility analysis.

Table 1: Child-Pugh classification of liver function

* Score 1 2 3

  * Ascites Absent Slight to moderate Severe
  * Encephalopathy Absent Slight to moderate Severe
  * Serum albumin >3.5 g/dl 3-3.5 g/dl <3 g/dl
  * Serum bilirubin <2 mg/dl 2-3 mg/dl >3 mg/dl
  * Prolongation of prothrombin time <4 seconds 4-6 seconds >6 seconds
* Score of 5 to 6 corresponds to Child-Pugh class A
* Score of 7 to 11 corresponds to Child-Pugh class B
* Score of 12 to 15 corresponds to Child-Pugh class
* The effects of gemcitabine+cisplatin on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study treatment. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately. Female patients of child bearing potential must indicate to their physician that they are not pregnant at the time of enrollment or have a negative serum pregnancy test.
* Ability to understand and the willingness to sign a written informed consent document.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Participants who exhibit any of the following conditions at screening will not be eligible for admission into the study.
* Participants who have had chemotherapy or radiotherapy for intrahepatic cholangiocarcinoma.
* Participants receiving any other anti-cancer or investigational agents.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to gemcitabine or cisplatin.
* Women who are pregnant or lactating.
* Participants with evidence of non-hepatic metastatic disease.
* Local conditions or systemic illnesses which would reduce the local tolerance to radiation treatment, such as serious local injuries, active collagen vascular disease, etc.
* Participants with a serious medical illness which may limit expected survival to less than 3 months.
* Participants with serious psychiatric illness or social situations which would limit adherence to study requirements.
* Participants receiving any medications or substances that are strong inhibitors or inducers of CYP3A4 are ineligible.
* Because no dosing or adverse event data are currently available on the use of gemcitabine+cisplatin in participants <18 years of age, children are excluded from this study.
* Patients who require anticoagulation should receive low-molecular weight or standard heparin and not warfarin.
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because gemcitabine is a class D agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk of adverse events in nursing infants secondary to treatment of the mother with gemcitabine, breastfeeding should be discontinued if the mother is treated with gemcitabine. These potential risks may also apply to other agents used in this study.
* Individuals with a history of a different malignancy are ineligible except for the following circumstances. Individuals with a history of other malignancies are eligible if they have been disease-free for at least 5 years and are deemed by the investigator to be at low risk for recurrence of that malignancy. Individuals with the following cancers are eligible if diagnosed and treated within the past 5 years: cervical cancer in situ, DCIS, stage I prostate cancer, and basal cell or squamous cell carcinoma of the skin.
* HIV-positive individuals on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with gemcitabine+cisplatin. In addition, these individuals are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in participants receiving combination antiretroviral therapy when indicated. HIV-positive individuals on HAART will be considered eligible of they have demonstrated good compliance and have a CD4 count > 500.
* Prior liver directed radiation.
* Patients with peripheral neuropathy ≥ grade 2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2014-10; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Theodore S. Hong, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 3 patients were enrolled between November 2014 and July 2015.
Groups:
- Resectable Disease: * Consent and Registration
  * 3 cycles of gemcitabine + cisplatin
  * Evaluate for surgery* (weeks 10-15)
    -- Patients who are eligible for surgery at restaging will receive surgery; patients not eligible for surgery at restaging will receive radiation therapy.
  * Proceed to surgery
  * Additional care as recommended; may include additional cycles of GEM + CDDP on a 21 day cycle and/or post-op radiation as recommended by treating medical oncologist and radiation oncologist
  Gemcitabine
  Cisplatin
  Surgery: Surgical Resection and Lymphadenectomy
- Unresectable Disease: * Consent and Registration
  * 3 cycles of gemcitabine + cisplatin
  * Evaluate for surgery* (weeks 10-15)
  * Patients who are eligible for surgery at restaging will receive surgery; patients not eligible for surgery at restaging will receive radiation therapy.
  * Proceed to radiation therapy with protons or photons, determined by available resources
  * Additional cycles of GEM + CDDP on a 21 day cycle as recommended by treating medical oncologist
  Gemcitabine
  Cisplatin
  Radiation: Radiation Therapy
Period: Overall Study
Arm/Group | Resectable Disease | Unresectable Disease
Started | 1 | 2
Completed | 1 | 1
Not Completed | 0 | 1
Not completed — Disease Progression | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Resectable Disease | Unresectable Disease | Total
Number analyzed (Participants) | 1 | 2 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 2 | 2
  >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Post Operative/Radiation Therapy Complications
Description: Out of the 3 participants enrolled, the patient in cohort 1 proceeded to surgery and 1 of the 2 patients in cohort 2 proceeded to RT. The other patient in cohort 2 developed disease progression and was removed from protocol.
Time Frame: 90 Days
Measure: Number; unit: participants
Arm/Group | Resectable Disease | Unresectable Disease
Number analyzed (Participants) | 1 | 1
participants | 0 | 0

ADVERSE EVENTS:
Arm/Group | Resectable Disease | Unresectable Disease
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/2
Other Adverse Events (participants affected / at risk) | 0/1 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes